CLINICAL TRIAL: NCT00296647
Title: Tobacco Dependence: Treatment and Outcomes; Pharmacotherapies: Effectiveness in Primary Care
Brief Title: Smoking Cessation Intervention: Effectiveness in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2004-0462; P50DA019706 (NIH); NCT00106873 (obsolete NCT alias)
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Bupropion; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- patch (Active Comparator)
  Interventions: Drug: nicotine patch
- nicotine lozenge (Active Comparator)
  Interventions: Drug: nicotine lozenge
- bupropion (Active Comparator)
  Interventions: Drug: bupropion
- patch + lozenge (Active Comparator)
  Interventions: Drug: patch + lozenge
- buproion + lozenge (Active Comparator)
  Interventions: Drug: bupropion + lozenge

INTERVENTIONS:
Drug: nicotine patch — Decreasing dosages from 21 to 7 mg over 12 week period
  Arms: patch
Drug: nicotine patch — Decreasing dosage from 21 to 7 mg over 12 weeks
  Arms: patch
Drug: nicotine lozenge — 4 mg nicotine lozenge: dosage according to package directions for 16 weeks
  Arms: nicotine lozenge
Drug: bupropion — dosage according to prescription directions: 12 weeks
  Arms: bupropion
Drug: patch + lozenge — dosage of each according to package insert directions (12 weeks patch, 16 weeks lozenge)
  Arms: patch + lozenge
Drug: bupropion + lozenge — dosage of each according to prescription or package insert (12 weeks bupropion, 16 weeks lozenge)
  Arms: buproion + lozenge

SUMMARY:
The information gathered in this study may help to develop more effective ways to help people quit smoking and stay quit in the future.

DETAILED DESCRIPTION:
Randomized clinical trials may not accurately reflect the public health benefit of tobacco dependence pharmacotherapies when used in real-world clinical settings due to differences in patient selection, motivation, and adherence. To have a positive public health impact, a treatment must be accessible and acceptable to a broad range of smokers and effective under normal use conditions. The proposed project will assess primary care patients willingness to use cessation treatment and will determine the relative effectiveness of five cessation pharmacotherapies. This research builds on a primary care clinic-based recruitment strategy that was highly successful in a previous study. In the proposed research, 1320 primary care patients presenting for a regular outpatient visit will be recruited by medical assistants to participate in a free smoking cessation program and will be randomly assigned to one of five active pharmacotherapies: patch, lozenge, bupropion, patch+lozenge, and bupropion+lozenge (n = 264/condition). Interested participants who pass medical screening will pick up their medications at clinic pharmacies and will receive proactive telephone counseling from the Wisconsin Tobacco Quit Line. Assessment will be limited to preserve the generalizability of the findings, but select individual differences will be assessed pre-quit to validate algorithms (from Project 1: Efficacy) designed to optimize pharmacotherapy selection for smokers based on gender, level of dependence, and other factors. Smoking behavior will be assessed at six months and one year post-quit so that abstinence rates across pharmacotherapy conditions can be compared. The cost of incorporating tobacco dependence treatment into primary care will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 10 cigarettes per day for the previous 6 months - Expired CO > 9 ppm - Motivated to quit smoking - Able to read and write English - Willing to complete required study assessments, Aurora participating clinic patient

Exclusion Criteria:

* Uncontrolled hypertension (systolic >180mm Hg or diastolic >110mm Hg) - History of bipolar disorder or psychosis - Myocardial infarction or other serious cardiac problem in the previous 4 weeks - History of diagnosed anorexia and/or bulimia - Diagnosis of Alcohol Dependence in the previous 6 months by participant self-report or drinking 6 or more drinks on six or more days a week - History of seizure and/or serious head injury involving loss of consciousness - Use of contraindicated medications (MAO inhibitors, bupropion, lithium, anticonvulsants, antipsychotics) - Currently pregnant or breast-feeding - Unwilling to use effective contraception during the treatment phase - More than one participant from the same household - Allergic reactions to 3 or more classes of drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1346 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Jackson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- UW-CTRI Milwaukee Research site, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Hockenberry JM, Curry SJ, Fishman PA, Baker TB, Fraser DL, Cisler RA, Jackson TC, Fiore MC. Healthcare costs around the time of smoking cessation. Am J Prev Med. 2012 Jun;42(6):596-601. doi: 10.1016/j.amepre.2012.02.019. PMID 22608375
- [Derived] Smith SS, McCarthy DE, Japuntich SJ, Christiansen B, Piper ME, Jorenby DE, Fraser DL, Fiore MC, Baker TB, Jackson TC. Comparative effectiveness of 5 smoking cessation pharmacotherapies in primary care clinics. Arch Intern Med. 2009 Dec 14;169(22):2148-55. doi: 10.1001/archinternmed.2009.426. PMID 20008701
- See also: web site of the study lead investigators — http://www.ctri.wisc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 1346 smokers recruited in 12 Aurora Health Care primary care clinics in eastern Wisconsin from October 2005 through May 2007.
Pre-assignment Details: Primary inclusion criteria included (1) 18 years or older; (2) 10 or more cigarettes per day (CPD) for the past 6 months; (3) motivated to quit smoking; and (4) if female, willing to use an acceptable contraception while using the study medication.
Period: Overall Study
Arm/Group | Patch | Nicotine Lozenge | Bupropion | Patch + Lozenge | Buproion + Lozenge
Started | 282 | 261 | 256 | 279 | 268
Completed | 250 | 233 | 222 | 262 | 248
Not Completed | 32 | 28 | 34 | 17 | 20
Not completed — Death | 4 | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 28 | 27 | 32 | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patch | Nicotine Lozenge | Bupropion | Patch + Lozenge | Buproion + Lozenge | Total
Number analyzed (Participants) | 282 | 261 | 256 | 279 | 268 | 1346
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.4) | 42.9 (11.7) | 44 (11.6) | 44.8 (12.4) | 45.4 (12.2) | 44.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 142 | 143 | 158 | 152 | 753
  Male | 124 | 119 | 113 | 121 | 116 | 593
Region of Enrollment [Number; unit: participants]
  United States | 282 | 261 | 256 | 279 | 268 | 1346

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Self-reported Abstinence From Smoking
Description: Primary postquit outcomes was 7-day point prevalence abstinence (0, abstinent; 1, smoking) at 6 months (based on the week 24 interview)
Time Frame: 6 months
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | Patch | Lozenge | Bupropion | Patch + Lozenge | Buproion + Lozenge
Number analyzed (Participants) | 279 | 261 | 256 | 279 | 268
participants | 50 | 52 | 45 | 75 | 80

ADVERSE EVENTS:
Time Frame: 6 months collection at scheduled follow up time points
Arm/Group | Patch | Nicotine Lozenge | Bupropion | Patch + Lozenge | Buproion + Lozenge
Serious Adverse Events (participants affected / at risk) | 4/282 | 1/261 | 2/256 | 1/279 | 1/268
Other Adverse Events (participants affected / at risk) | 18/282 | 15/261 | 12/256 | 13/279 | 6/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patch (N=282) | Nicotine Lozenge (N=261) | Bupropion (N=256) | Patch + Lozenge (N=279) | Buproion + Lozenge (N=268)
death (Cardiac disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patch (N=282) | Nicotine Lozenge (N=261) | Bupropion (N=256) | Patch + Lozenge (N=279) | Buproion + Lozenge (N=268)
skin irritation (Skin and subcutaneous tissue disorders) | 15 (15) | 3 (3) | 6 (6) | 5 (5) | 3 (3)
nausea (Gastrointestinal disorders) | 3 (3) | 12 (12) | 6 (6) | 8 (8) | 3 (3)

LIMITATIONS AND CAVEATS:
The present study is limited to some extent by the fact that self-reported abstinence was not biochemically confirmed. However, there is evidence that self-reported abstinence rates are generally accurate in low-contact effectiveness studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No